CLINICAL TRIAL: NCT02277067
Title: Carbetocin Versus Misoprostol for Prevention of Postpartum Hemorrhage in Pregnant Women at High Risk Following C.S.
Brief Title: Carbetocin Versus Misoprostol in High Risk Patients for Postpartum Hemorrhage After C.S.
Acronym: PPH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Nesreen Abdel Fattah Abdullah Shehata, Lecturer of Obstetrics and Gynecology, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Beni-Suef 7
Record Dates: First submitted 2014-10-26; First posted 2014-10-28 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Postpartum Hemorrhage
Keywords: PPH
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — carbetocin; Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pabal ( carbetocin) (Active Comparator): Pabal (carbetocin which is a long acting oxytocin ) given as 100 mcg slow i.v. injection over 1 minute ( Draxis/Multiph). It will be given to the patients included in the study after delivery of the fetal head.
  Interventions: Drug: Carbetocin
- Misoprostol (Active Comparator): Misoprostol ( Misotac, Sigma, Egypt) is a stable, synthetic form of prostaglandin E1 analogue. Patients wil be given 600 microgram of misotac immediately postoperative.
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Carbetocin — Pabal 100 mcg iv infusion over 1 minute given after delivery of fetal head In the first group of patients, carbitocin 100 mcg will be given iv infusion over one minute after delivery of the head in cesarean section.
  Other Names: Pabal
  Arms: Pabal ( carbetocin)
Drug: Misoprostol — 600 micro gram of misoprostol which is a prostaglandin E1 will be given per rectum for patients immediately postoperative.
  Other Names: Misotac
  Arms: Misoprostol

SUMMARY:
We will compare between Carbitocin and Misoprostol in prevention of postpartum hemorrhage in high risk patients after C.S.

DETAILED DESCRIPTION:
* Postpartum hemorrhage was traditionally defined as blood loss in excess of 500 mL from a vaginal delivery or 1000 mL at cesarean section. It can result from uterine atony, retained placental tissue including that from abnormal placentation, maternal genital tract trauma and coagulopathies. (Almog et al, 2011)
* Uterotonic agents (e.g. ergometrine, misoprostol) should be easily accessible. Many units of an oxytocin infusion and/or rectal misoprostol during and after cesarean deliveries used to reduce the incidence of atony. -Misoprostol has been widely recommended for the prevention of post-partum hemorrhage when other methods are not available. The most common regimen reported for the treatment of post-partum hemorrhage is rectally. (Oladapo et al., 2012)
* Misoprostol is a prostaglandin E1 analogue. It has been investigated in the prevention of postpartum hemorrhage, using either the oral or rectal route of administration. (Hofmeyr et al, 2009)
* Carbetocin is a long-acting oxytocin studied by Dansereau et al.; 1999.They found that the carbetocin group of patients had a decreased incidence of PPH and of the need for therapeutic oxytocics. The recommended dose of carbetocin is 100 mg given either IM or slowly (over 1 minute).
* Risk factors may present antenatally or intrapartum; care plans must be modified when risk factors present. Clinicians must be aware of risk factors for PPH and should take these into account for the wellbeing and safety of both the mother and the baby.RCOG GUIDLIN Table 1: Risk factors for PPH

  * Suspected or proven placental abruption
  * Known placenta praevia
  * Multiple pregnancy
  * Pre-eclampsia/gestational hypertension
  * Previous PPH .
  * Obesity (BMI >35)
  * Anaemia (<9 g/dl)
  * Delivery by elective caesarean section
  * Induction of labour
  * Retained placenta Tissue
  * Prolonged labour (> 12 hours) .
  * Big baby (> 4 kg) Royal College of Obstetrics and Gynecology.Green-top Guideline No. 52 May 2009 Minor revisions November 2009 and April 2011. Prevention and Management of Postpartum Hemorrhage. Thus our aim is to compare the effeciency and cost effectiveness of Carbitocin and Misoprostol in patients at high risk of PPH after C.S. in prevention of PPH.

ELIGIBILITY:
Inclusion Criteria:

* Women with a singleton pregnancy undergoing cesarean section after 37 weeks of gestation.

Any medical disorder with pregnancy that carries a risk factor for PPH.

Exclusion Criteria:

* Women undergoing cesarean section with general anesthesia will be excluded, because carbetocin is licensed for use with regional anaesthesia only.
* women undergoing cesarean section at less than 37 weeks of gestation.

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-10; Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Uterine tone and size | One hour after the cesarean section
  The uterine tone and size will be assessed by using a hand resting on the fundus and palpating the anterior wall of the uterus one hour after the operation. The presence of a boggy uterus with either heavy vaginal bleeding or increasing uterine size can suspect diagnosis of uterine atony.

SECONDARY OUTCOMES:
Blood loss | One hour after cesarean section
  Blood loss will be estimated postoperatively by giving each woman of each group standard 2 dressings (standard weight of dressing is 25 gm) for one hour postoperative and recording weight of blood soaked dressings and volume of lost blood.

OTHER OUTCOMES:
Hemoglobin concentration | Before and 24 hours after the operation
  Changes in hemoglobin concentrations before and 24 hours postoperative. Using a 10% fall in hematocrit value to define post-partum hemorrhage.

CONTACTS AND LOCATIONS:
Overall Officials: Nesreen A Shehata, MD, Principal Investigator — Beni-Suef University
Locations (1):
- Beni-Suef University, Cairo, Egypt

REFERENCES:
- See also: • Almog B,Malabarey O, Brown R, Abenhaim HA, Shrim A. (2011), Postpartum hemorrhage in low risk population. J Perinat Med. 2011 Sep; 39(5):495-8. Epub 2011 Jun 30. Department of Obstetrics and Gynecology, McGill University Health Center, Montreal, QC, — http://www.google.com.eg/webhp?sourceid=chrome-instant&ion=1&espv=2&ie=UTF-8#q=%E2%80%A2%20Almog%20B%2CMalabarey
- See also: Advance misoprostol distribution for preventing and treating postpartum haemorrhage. Cochrane Database Syst Rev. 2012 Feb 15; 2:CD009336. Maternal and Fetal Health Research Unit, Department of Obstetrics and Gynaecology, Obafemi Awolowo College of Health — http://www.google.com.eg/webhp?sourceid=chrome-instant&ion=1&espv=2&ie=UTF-8#q=Oladapo%20et%20al.%2C%202012)
- See also: Maternal consequences of caesarean section. A retrospective study of intra-operative and postoperative maternal complications of caesarean section during a 10- year period. Eur J Obstet Gynecol Reprod Biol. 2009;74(1):1-6. — http://www.google.com.eg/webhp?sourceid=chrome-instant&ion=1&espv=2&ie=UTF-8#q=Hofmeyr+et+al%2C+2009
- See also: • Dansereau J, Joshi AK, Helewa ME, Doran TA, Lange IR, Luther ER, et al. Double-blind comparison of carbetocin versus oxytocin in prevention of uterine atony after cesarean section. Am J Obstet Gynecol 1999; 180:670-6. — http://www.google.com.eg/webhp?sourceid=chrome-instant&ion=1&espv=2&ie=UTF-8#q=Dansereau+et+al.%3B+1999